CLINICAL TRIAL: NCT03609294
Title: A Randomized, Open-label, Single Dose, 3x3 Partial Replicated Crossover Study to Evaluate the Pharmacokinetics and Safety/Tolerability Between a Fixed Dose Combination of Fimasartan 120 mg/Linagliptin 5 mg and Co-administration of Fimasartan 120 mg and Linagliptin 5 mg in Healthy Male Volunteers
Brief Title: A Clinical Trial to Evaluate the Pharmacokinetics and Safety/Tolerability of Fimasartan and Linagliptin in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BR-FLC-CT-102
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Hypertension; Diabetes
Keywords: Fimasartan; Linagliptin
MeSH Terms: conditions — Hypertension; Diabetes Mellitus | interventions — fimasartan; Linagliptin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sequence A (Experimental): Period 1(Treatment A) - Period 2(Treatment A) - Period 3(Treatment B)
  There will be a washout of 35 days between the each period.
  Interventions: Drug: Treatment A (Fimasartan, Linagliptin); Drug: Treatment B (Fimasartan/Linagliptin)
- Sequence B (Experimental): Period 1(Treatment A) - Period 2(Treatment B) - Period 3(Treatment A)
  There will be a washout of 35 days between the each period.
  Interventions: Drug: Treatment A (Fimasartan, Linagliptin); Drug: Treatment B (Fimasartan/Linagliptin)
- Sequency C (Experimental): Period 1(Treatment B) - Period 2(Treatment A) - Period 3(Treatment A)
  There will be a washout of 35 days between the each period.
  Interventions: Drug: Treatment A (Fimasartan, Linagliptin); Drug: Treatment B (Fimasartan/Linagliptin)

INTERVENTIONS:
Drug: Treatment A (Fimasartan, Linagliptin) — Co-administration of Fimasartan and Linagliptin
Drug: Treatment B (Fimasartan/Linagliptin) — Fixed Dose Combination of Fimasartan 120 mg/Linagliptin 5 mg

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety/tolerability when administrated fixed dose combination of Fimasartan/Linagliptin and when co-administrated Fimasartan and Linagliptin.

DETAILED DESCRIPTION:
This is an open-label, randomized, 3x3 partial replicated crossover study to evaluate the pharmacokinetics and safety/tolerability. Within each period, randomized subjects will be 2 dosing regimens with a fixed dose combination of Fimasartan/Linagliptin and co-administration of Fimasartan and Linagliptin.

ELIGIBILITY:
Inclusion Criteria:

1. Male 19-50 years of age.
2. Body mass index (BMI) ≥ 18 and ≤ 27 kg/m2 at screening.
3. Understands the study procedures in the Informed consent form (ICF), and be willing and able to comply with the protocol.
4. Medically healthy with no clinically significant medical history.

Exclusion Criteria:

1. History or presence of clinically significant medical or psychiatric condition or disease.
2. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
3. Seated blood pressure is less than 100/55 mmHg or greater than 140/100 mmHg at screening.
4. Plasma donation within a month prior to the first dose of study drug.
5. Participation in another clinical trial within 3 months prior to the first dose of study drug(s).

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-03-04 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Cmax | Fimasartan: 0-48 hours after administration, Linagliptin: 0-72 hours after administration
  Maximum concentration of drug in plasma of Fimasartan, Linagliptin
AUClast | Fimasartan: 0-48 hours after administration, Linagliptin: 0-72 hours after administration
  Area under the plasma drug concentration-time curve over the time interval from 0 to the last observed plasma concentration of Fimasartan, Linagliptin

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Sang Yu, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Dahak-ro, South Korea

IPD SHARING:
Plan to Share IPD: No